CLINICAL TRIAL: NCT01341509
Title: Insertional Achilles Tendinopathy: A Randomized Trial to Evaluate the Effectiveness of Transferring the Flexor Hallucis Longus Tendon
Brief Title: A Randomized Trial to Evaluate the Effectiveness of Transferring the Flexor Hallucis Longus Tendon
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: OAD Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GW100
Record Dates: First submitted 2011-04-22; First posted 2011-04-25 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Achilles Tendinopathy
Keywords: Surgical Treatment of Insertional Achilles Tendinopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- FHL tendon transferred (Active Comparator): Surgical group in which the FHL tendon was transferred
  Interventions: Procedure: Transfer of the Flexor Hallucis Longus Tendon
- FHL tendon not transferred (Active Comparator)
  Interventions: Procedure: Flexor Hallucis Longus Tendon transfer; Procedure: No transfer of Flexor Hallucis Longus tendon

INTERVENTIONS:
Procedure: Flexor Hallucis Longus Tendon transfer — The flexor hallucis longus tendon was transferred during surgery for insertional achilles tendinopathy
  Arms: FHL tendon not transferred
Procedure: Transfer of the Flexor Hallucis Longus Tendon — The Flexor Hallucis Longus Tendon was transferred during surgery for insertional achilles tendinopathy
  Arms: FHL tendon transferred
Procedure: No transfer of Flexor Hallucis Longus tendon — There was no transfer of the Flexor Hallucis Longus tendon in surgery for insertional achilles tendinopathy
  Arms: FHL tendon not transferred

SUMMARY:
The optimal surgical treatment for insertional Achilles tendinopathy remains unclear. The purpose of this study is to evaluate the long-term outcome of surgical treatment by comparing the patient reported outcomes of Insertional Achilles Tendinopathy; Achilles tendon debridement, excision calcaneal exostosis, Strayer procedure, secondary repair of Achilles with flexor hallucis longus (FHL) transfer and Achilles tendon debridement, excision calcaneal exostosis, Strayer procedure, secondary repair of Achilles without FHL transfer.

ELIGIBILITY:
Inclusion Criteria:

* Male and female 18 years or older
* Diagnosed with insertional Achilles tendinosis by history and physical exam
* Confirmed by x-ray and MRI
* Calcification at the Achilles insertion and gastrocnemius tightness.
* Failure of the following non-operative treatment for greater than 6 months: *shoe modifications

  * physical therapy
  * immobilization
  * and home exercise program.
* In addition, participant must have an intact flexor hallucis longus tendon.

Exclusion Criteria:

* Patients who have failed surgery for the same and patients with diabetic neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Statistical difference | 2 years
  To detect a 20% difference in clinical outcomes between the two surgical groups.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory P Witkowski, MD, Principal Investigator — OAD Orthopaedics
Locations (1):
- OAD Orthopaedics, Warrenville, Illinois, United States